CLINICAL TRIAL: NCT04601506
Title: PRescribing INterventions for Chronic Pain Via the Electronic Health Record Study - Primary Care Providers
Acronym: PRINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006522-3; R33DA046084 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Opioid-use Disorder; Opioid Use; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: 43 Primary Care Clinics will be randomized to be in one of 4 arms: 1) Care as usual, 2) Choice architecture nudge, 3) Prescription Drug Monitoring Program (PMP) Integration & nudge, 4) Choice architecture nudge + PMP Integration & nudge
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Care as Usual (No Intervention): Clinics assigned to this arm will continue to care for the patients as usual in regards to opioid prescribing.
- Choice Architecture Nudge (Experimental): Clinics in this arm will receive the choice architecture nudge intervention.
  Interventions: Behavioral: Choice Architecture Nudge
- PMP Integration & Nudge (Experimental): Clinics in this arm will receive the Prescription Drug Monitoring (PMP) Integration & Nudge intervention.
  Interventions: Behavioral: PMP Integration & Nudge
- Choice Architecture Nudge + PMP Integration & Nudge (Experimental): Clinics in this arm will receive both the choice architecture nudge and prescription drug monitoring (PMP) integration & nudge interventions.
  Interventions: Behavioral: Choice Architecture Nudge; Behavioral: PMP Integration & Nudge

INTERVENTIONS:
Behavioral: Choice Architecture Nudge — Primary Care Providers (PCPs) will be sent alerts in the Electronic Health Record system when they initiate an opioid order for a patient who has not had an opioid prescription within the past six months. The alert provides guidance language about opioid prescribing and prompts the PCP to open the "SmartSet" to order non-opioid treatment alternatives. When the SmartSet is opened, PCPs can choose to click on a variety of treatment order options, including both non-opioid pharmacological options and non-pharmacological options.
  PCPs will also be sent alerts when they initiate an opioid order for a patient will a current opioid prescription. The alerts prompt PCPs to consider tapering the patient's opioid. The alert also displays the MME of the patient's current opioid prescription and automatically calculates what a 10% reduction in MME relative to the current prescription would be. The alert contains options to either cancel the refill order, or to continue with the order.
  Arms: Choice Architecture Nudge; Choice Architecture Nudge + PMP Integration & Nudge
Behavioral: PMP Integration & Nudge — During the Prescription Drug Monitoring Program (PMP) integration & nudge intervention, Primary Care Providers (PCPs) will have integrated access to the PMP embedded within the EHR. All clinicians can already access the PMP to look up a patient's prior opioid prescriptions and prescription fills. However, this process involves signing in to the separate PMP website and can be complicated and time-consuming within typical clinical workflow. The integrated PMP tool makes it much easier and faster for a PCP to access the PMP information for a given patient.
  Arms: Choice Architecture Nudge + PMP Integration & Nudge; PMP Integration & Nudge

SUMMARY:
The objective of this research is to assess the effects of electronic health record (EHR)-based decision support tools on primary care provider (PCP) decision-making around pain treatment and opioid prescribing. The decision support tools are informed by principles of "behavioral economics," whereby clinicians are "nudged," though never forced, towards guideline-concordant care.

DETAILED DESCRIPTION:
To test the effects of these decision support tools for improving the quality of care for pain treatment, the investigators will implement a pragmatic clinic-randomized trial across the primary care clinics of Fairview Medical Group and University of Minnesota Physicians.

The study has two parallel components. The decision support tools to be tested will differ somewhat depending on whether a given patient is opioid-naïve, or whether a given patient is a current opioid-user. Four sets of analyses will be conducted separately: one for the opioid-naïve group using EHR data, one for the current opioid-user group using EHR data, one at the PCP-level using web survey data, and one at the PCP-level using MN Prescription Drug Monitoring Program (PDMP) data.

ELIGIBILITY:
Inclusion Criteria:

- All primary care providers from all of the Fairview and University of Minnesota Physicians study clinics

Exclusion Criteria:

- Primary care providers who work less than 20% full time equivalent (FTE)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Golberstein, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Neprash HT, Vock DM, Hanson A, Elert B, Short S, Karaca-Mandic P, Rothman AJ, Melton GB, Satin D, Markowitz R, Golberstein E. Effect of Integrating Access to a Prescription Drug Monitoring Program Within the Electronic Health Record on the Frequency of Queries by Primary Care Clinicians: A Cluster Randomized Clinical Trial. JAMA Health Forum. 2022 Jun 5;3(6):e221852. doi: 10.1001/jamahealthforum.2022.1852. eCollection 2022 Jun. PMID 35977248

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original study protocol included a potential second randomization period after six months into the trial. This secondary randomization did not occur, per the recommendation of the Data Monitoring Committee
Units Other Than Participants: clinics
Groups:
- Choice Architecture Nudge: Clinics in this arm will receive the choice architecture nudge intervention.
  Choice Architecture Nudge: Primary Care Providers (PCPs) will be sent alerts in the Electronic Health Record system when they initiate an opioid order for a patient who has not had an opioid prescription within the past six months. The alert provides guidance language about opioid prescribing and prompts the PCP to open the "SmartSet" to order non-opioid treatment alternatives. When the SmartSet is opened, PCPs can choose to click on a variety of treatment order options, including both non-opioid pharmacological options and non-pharmacological options.
  PCPs will also be sent alerts when they initiate an opioid order for a patient will a current opioid prescription. The alerts prompt PCPs to consider tapering the patient's opioid. The alert also displays the MME of the patient's current opioid prescription and automatically calculates what a 10% reduction in MME relative to the current prescription would be. The alert contains options to either cancel the refill order, or to continue with the order.
- Choice Architecture Nudge + PMP Integration & Nudge: Clinics in this arm will receive both the choice architecture nudge and prescription drug monitoring (PMP) integration & nudge interventions.
  Choice Architecture Nudge: Primary Care Providers (PCPs) will be sent alerts in the Electronic Health Record system when they initiate an opioid order for a patient who has not had an opioid prescription within the past six months. The alert provides guidance and prompts open the "SmartSet" to order non-opioid treatment alternatives.
  PCPs will also be sent alerts when they initiate an opioid order for a patient will a current opioid prescription. The alerts prompt PCPs to consider tapering the patient's opioid. The alert also displays the MME of the patient's current opioid prescription and automatically calculates what a 10% reduction in MME relative to the current prescription would be.
  PMP Integration & Nudge: During the Prescription Drug Monitoring Program (PMP) integration & nudge intervention, Primary Care Providers (PCPs) will have integrated access to the PMP embedded within the EHR. All clinicians can already access the PMP to look up a patient's prior opioid prescriptions and prescription fills. However, this process involves signing in to the separate PMP website and can be complicated and time-consuming within typical clinical workflow. The integrated PMP tool makes it much easier and faster for a PCP to access the PMP information for a given patient.
Period: Overall Study
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Started | 79; 11 clinics | 69; 11 clinics | 74; 10 clinics | 87; 11 clinics
Completed | 79; 11 clinics | 69; 11 clinics | 74; 10 clinics | 87; 11 clinics
Not Completed | 0; 0 clinics | 0; 0 clinics | 0; 0 clinics | 0; 0 clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge | Total
Number analyzed (Participants) | 79 | 69 | 74 | 87 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] — Age information was not collected Population: Age information not collected
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 39 | 42 | 40 | 59 | 180
  Male | 36 | 25 | 32 | 27 | 120
  Unknown | 4 | 2 | 2 | 1 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequency of PDMP Checks
Description: Outcome is reported as the mean number of times an individual Primary Care Provider checks the Prescription Drug Monitoring Program per month.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: PDMP queries per PCP per month
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Number analyzed (Participants) | 79 | 69 | 74 | 87
PDMP queries per PCP per month | 19 (89.2) | 23 (28.2) | 31.9 (26.7) | 22.1 (32.3)

2. Secondary Outcome: PCP Satisfaction #1
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (very unsatisfied) to 5 (very satisfied): "How would you rate your overall satisfaction with the best practice (BPA) alerts (pop-ups) and clinical decision support you received in the EHR for opioid prescribing for patients with acute pain?"
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: PCP Satisfaction #2
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (very unsatisfied) to 5 (very satisfied): "How would you rate your overall satisfaction with the best practice (BPA) alerts (pop-ups) and clinical decision support you received in the EHR for opioid prescribing for patients with chronic pain?"
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: PCP Satisfaction #3
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (very unsatisfied) to 5 (very satisfied): "How would you rate your overall satisfaction with the PDMP when prescribing opioids for patients with acute pain?"
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: PCP Satisfaction #4
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (very unsatisfied) to 5 (very satisfied): "How would you rate your overall satisfaction with the PDMP when prescribing opioids for patients with chronic pain?"
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: PCP Satisfaction #5
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (very easy) to 5 (very difficult): "Over the past year, how easy or difficult was it to access information on prescription drug use for your own patients in the PDMP?"
Time Frame: 12 months
Reporting Status: Not Posted

7. Secondary Outcome: PCP Satisfaction #6
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (not useful at all) to 5 (very useful): "Over the past year, how useful was the information that you accessed from the PDMP?"
Time Frame: 12 months
Reporting Status: Not Posted

8. Secondary Outcome: PCP Satisfaction #7
Description: In order to assess satisfaction with the electronic health record-based decision support tools, Primary Care Providers (PCP) will be asked to answer the following question on a scale from 1 (a lot more) to 5 (a lot less): "Compared to 12 months ago, how frequently are you engaging patients in discussions about opioids?"
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events not collected
Description: Adverse events not collected
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT04601506/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04601506/ICF_001.pdf